CLINICAL TRIAL: NCT03822169
Title: Choline Uptake Study
Acronym: CUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: AAK (Other)
Responsible Party: Principal Investigator, Diederik Esser, project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NL67054.081.18
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Choline Uptake; Kinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline added as a phospholipid (Experimental): A shake with phospholipid-bound choline (and bound DHA),
  Interventions: Dietary Supplement: Choline added as a phospholipid
- Choline added as a salt (Active Comparator): control shake with choline added as a salt and added DHA.
  Interventions: Dietary Supplement: Choline added as a salt

INTERVENTIONS:
Dietary Supplement: Choline added as a phospholipid — A shake with 3000 mg choline added as a phospholipid
  Arms: Choline added as a phospholipid
Dietary Supplement: Choline added as a salt — A shake with 3000 mg choline added as a salt
  Arms: Choline added as a salt

SUMMARY:
The study is a randomised, cross-over, double blind, controlled trial in which study participants will visit the research facility on two occasions under fasting conditions with a washout period of one week. During each visit, study subjects will receive a test shake with phospholipid-bound choline or a control shake with choline added as a salt and DHA added separately. The two shakes will be given in randomised order and blood will be collected via a catheter before and up-to 6 hours after choline consumption. All study participants will receive a standardised evening meal prior to each study day and asked not to drink alcohol or perform heavy exercise the day before each study day. Study subjects are also asked to avoid choline rich products the day before each test day. Study participants are offered a meal after the test day.

DETAILED DESCRIPTION:
Choline is water-soluble vitamin-like essential nutrient. It is made in small amounts by the liver, but humans need to receive choline through the diet or by supplementation for proper health. Pregnancy and lactation are times when demand for choline is especially high. Infant formula not made from cow's milk is therefore supplemented with choline. Choline is therefore widely used. It is normally added to food products as a salt. However, if choline is present in a natural form, bound to phospholipids, it may be more efficiently absorbed. Docosahexaenoic acids (DHA) are also bound to these phospholipids.

The primary objective is determine choline uptake and bioavailability after consumption of a test shake with phospholipid-bound choline (and DHA), and to compare this to a control shake with choline added as a salt (and DHA added as an oil). Secondary objective is to compare the uptake and bioavailability of DHA after the two shakes.

The study is a cross-over, double blind, controlled trial in which study participants will visit the research facility on two occasions under fasting conditions. Subjects will receive two different choline products in randomized order with a washout period of one week. Blood will be collected via a catheter before and up-to 6 hours after choline consumption.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women
* Age between 30 and 70 years
* Body mass index (BMI) between 18.5 and 24.9 kg/m2
* Having veins suitable for blood sampling via a catheter (judged by study nurse/ medical doctor)

Exclusion Criteria:

* Any metabolic, gastrointestinal, inflammatory or chronic disease (such as diabetes, anaemia, hepatitis, cardiovascular disease)
* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery
* Kidney dysfunction (self-reported)
* Use of medication that may influence the study results,
* such as laxatives, stomach protectors and drugs that can affect intestinal motility.
* Use of choline or fish oil supplements
* Reported slimming, medically prescribed or vegan diet
* Current smokers
* Alcohol intake ≥4 glasses of alcoholic beverages per day
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported)
* Abuse of illicit drugs
* Food allergies for products that we use in the study
* Participation in another clinical trial at the same time
* Being an employee of the department Consumer Science & Health group of Wageningen Food & Biobased Research and/or Human Nutrition and Health

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
change in plasma choline concentration | blood samples will be taken before and up to 6 hours after shake consumption
  postprandial test, determine choline in blood samples collected before and after a shake
change in plasma betaine concentration | blood samples will be taken before and up to 6 hours after shake consumption
  postprandial test, determine betaine in blood samples collected before and after a shake
change in plasma dimethylglycine concentration | blood samples will be taken before and up to 6 hours after shake consumption
  postprandial test, determine dimethylglycine in blood samples collected before and after a shake

SECONDARY OUTCOMES:
Change in plasma DHA concentration | blood samples will be taken before and up to 6 hours after shake consumption
  postprandial test, determine DHA in blood samples collected before and after a shake

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No